CLINICAL TRIAL: NCT05272657
Title: Low-Carbohydrate Diet Versus Mediterranean Diet as Treatment for Women With Polycystic Ovary Syndrome.
Brief Title: Low-Carb Versus Mediterranean Diet in PCOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pcos2typesofDiet
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
Keywords: microbiome; obesity; Mediterranean diet; low-carb diet
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity | interventions — Diet, Carbohydrate-Restricted; Diet, Mediterranean

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-carbohydrate diet (Experimental): subjects in this arm are given detailed instructions and coaching in following a low-carbohydrate diet.
  Interventions: Other: low-carbohydrate diet
- Mediterranean diet (Experimental): subjects in this arm are given detailed instructions and coaching in following a Mediterranean diet.
  Interventions: Other: Mediterranean diet

INTERVENTIONS:
Other: low-carbohydrate diet — subjects in this arm are given detailed instructions and coaching in following a low-carbohydrate diet.
  Arms: low-carbohydrate diet
Other: Mediterranean diet — subjects in this arm are given detailed instructions and coaching in following a Mediterranean diet.
  Arms: Mediterranean diet

SUMMARY:
This is a randomized controlled trial of two diets (low-carbohydrate and Mediterranean diet) in the treatment of women with polycystic ovary syndrome (PCOS). The trial assesses the effects of the two diets on clinical, metabolic and hormonal parameters, inflammatory markers and gut microbiota . This study is an interventional, randomized controlled trial, open-labeled.

DETAILED DESCRIPTION:
The study aims to clarify the impact of nutritional recommendations for women with polycystic ovary syndrome on clinical, metabolic and hormonal parameters, inflammatory markers and gut microbiota . Women with PCOS are randomized into 2 treatment groups: one group on a low-carbohydrate diet and the other on a Mediterranean diet. The adhearance to a prescribed diet will be controlled through food intake diaries using a mobile application with electronic reporting forms.

ELIGIBILITY:
Inclusion Criteria:

* Women with PCOS between the ages of 18-40 years and with a body mass index of less than or equal to 45.
* Fulfillment of at least two of the following three criteria for PCOS, adopted by the Rotterdam Consensus in 2003 (Rotterdam ESHRE / ASRM-Sponsored PCOS Consensus Workshop Group):

  * signs of hyperandrogenemia - clinical and / or biochemical (increase in the index of free androgens or total testosterone)
  * signs of chronic anovulation
  * ultrasound signs: the number of follicles in the ovary ≥ 20 and / or ovarian volume ≥ 10 ml in any ovary in the case of gynecological age 8 or more years after menarche.

Exclusion Criteria:

* The presence of hyperprolactinemia
* Cushing's syndrome
* Ongenital hyperplasia of the adrenal cortex
* Hypothyroidism
* Androgen-producing tumors
* Regular use of drugs and dietary supplements that affect the function of the ovaries
* Adrenal glands
* Metabolism of carbohydrates
* Lipids
* Microbiota composition during the 2 months preceding the study
* Pregnancy
* Lactation
* Significant comorbidities

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-03-30 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
1. Homeostasis Model Assessment for Insulin Resistance (HOMA-IR) index | 12 weeks
  Changes in HOMA-IR index (fasting insulin [mU/l] * fasting glucose [mmol/L]/22.5) after intervention
2. Free androgen index | 12 weeks
  Changes in free androgen index [ (total testosterone level / sex hormone binding globulin (SHBG) level) * 100].

SECONDARY OUTCOMES:
1. Total testosterone | 12 weeks
  Changes in total testosterone levels [nmol/L] in serum after intervention
2. Androstenedione | 12 weeks
  Changes in androstenedione levels in serum after intervention [ng/ml]
3. Anti-Müllerian hormone (AMH) | 12 weeks
  Changes in AMH levels in serum after intervention [ng/ml]
4. 17-Hydroxyprogesterone (17-OH-progesterone) | 12 weeks
  Changes in 17-OH-progesterone levels in serum after intervention [ng/ml]
5. Luteinizing hormone (LH) | 12 weeks
  Changes in LH levels in serum after intervention [mU/ml]
6. Follicle-stimulating hormone (FSH) | 12 weeks
  Changes in FSH levels in serum after intervention [mU/ml]
7. Insulin | 12 weeks
  Changes in insulin levels in serum as measured with a two-hour oral glucose tolerance test (75 mg glucose in 300 ml water, blood draws at 0 minutes, 60 min and 120 min) [mU/l]
8. Glucose | 12 weeks
  Changes in glucose levels in plasma as measured with a two-hour oral glucose tolerance test (75 mg glucose in 300 ml water, blood draws at 0 minutes, 60 min and 120 min) [mmol/L]
9. Matsuda index | 12 weeks
  Changes in matsuda index after intervention measured with the formula M=10000/squareroot(glucose0 * insulin0 * Mean OGTT glucose concentration * Mean OGTT insulin concentration)
10. Hirsutism | 12 weeks
  measured by Ferriman-Gallwey-score (mFG-score), ranging from 0 to 36, with 0 being the best possible value and 36 the worst
11. Body-mass-index (BMI) | 12 weeks
  BMI measured with the formula BMI=weight [kg]/height² [m]
12. waist-to-hip ratio | 12 weeks
  Calculated with the formula: waist circumference/hip circumference
13. Gut microbiome composition | 12 weeks
  Changes in gut microbiome composition measured from stool samples via 16S-RNA gene sequencing
14. Inflammatory markers | 12 weeks
  Changes in inflammatory markers (Cytokines) measured by Human Cytokine/Chemokine/Growth Factor Panel A. 48 plex kit, pg/mL
15. Untargeted metabolomics | 12 weeks
  Serum samples will be analysed to identify biomarkers differentially changing in response to the studied diets using ultra-high performance liquid chromatography (UHPLC).
16. Untargeted metabolomics | 12 weeks
  Serum samples will be analysed to identify biomarkers differentially changing in response to the studied diets using ultra-high performance mass spectrometry (MS).
17. Serum Low-density lipoproteins (LDL) | 12 weeks
  Changes in serum Low-density lipoproteins (LDL), mmol/L
18. Serum high-density lipoproteins (LDL) | 12 weeks
  Changes in serum high-density lipoproteins (LDL), mmol/L
19. Serum triglyceride levels, mmol/L | 12 weeks
  Changes in serum triglyceride levels, mmol/L
20. Ovulation rate | 12 weeks
  Percent of women with ovulation recorded by serial transvaginal ultrasound after 8 weeks of participating in the study
21. Ovarian volume | 12 weeks
  Changes in ovarian volume (cm3) measured by transvaginal ultrasound in early follicular phase or after 3 months of amenorrhea

CONTACTS AND LOCATIONS:
Overall Officials: Polina Popova, MD,PhD, Study Chair — Almazov National Medical Research Centre

IPD SHARING:
Plan to Share IPD: No